CLINICAL TRIAL: NCT07096557
Title: Evaluation of the Effect of Co-enzyme Q10 on the Clinical Outcome of Pediatric Patients With Systemic Lupus Erythematosus
Brief Title: The Effect of Co-enzyme Q10 on the Clinical Outcome of Pediatric Patients With Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Helal, Demonstrator of clinical pharmacy department at faculty of pharmacy Ain shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2020110301 REC #272
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — coenzyme Q10

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Coenzyme Q10 group (Experimental): Group 1 (Coenzyme Q10 group): consists of 30 patients who will receive one capsule containing 100 mg Coenzyme Q10 once daily for 12 weeks, "Coenzyme Q10 Forte® ".
  Interventions: Drug: Coenzyme Q10
- Control group (No Intervention): Group 2 (Control group): consists of 30 patients who will not receive the intervention.

INTERVENTIONS:
Drug: Coenzyme Q10 — Coenzyme Q10 100 mg capsule once daily for 3 months
  Arms: Coenzyme Q10 group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of coenzyme Q10 supplementation in pediatric patients with SLE. The main questions it aims to answer are:

* What the impact of coenzyme Q10 supplementation on mitochondrial dysfunction?
* Does it have beneficial effect on disease activity through assessment of systemic lupus erythematosus disease activity index (SLEDAI) score?

Researchers will compare the group of patients that take coenzyme Q10 to a group that doesn't to see if coenzyme Q10 supplementation works to decrease mitochondrial dysfunction and disease activity.

Participants will:

Take coenzyme Q10 plus standard treatment of SLE or the standard treatment only every day for 3 months.

Visit the clinic once every 4 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders aged 6-16 years old diagnosed with SLE according to the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria of SLE.
2. Patients with moderate to severe activity presenting with lupus nephritis.
3. No enrollment in any other clinical trial.
4. Judged by the physician to be physically stable.

Exclusion Criteria:

1. Patients taking over-the-counter antioxidants such as N-acetylcysteine, vitamin E, omega-3 fatty acids, L-carnitine or vitamin C that can enhance the effect of CoQ10.
2. Patients with very severe active SLE that might threaten vital organs.
3. Patients with chronic infections, severe and recurrent infections whether bacterial, viral, or fungal infection

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial dysfunction | 3 months
  Through assessment of NLRP3 Inflammasome and Type 1 INF (INF α).

SECONDARY OUTCOMES:
systemic lupus erythematosus disease activity index (SLEDAI) score. | 3 months
  Determine its possible beneficial effect on disease activity through assessment of systemic lupus erythematosus disease activity index (SLEDAI) score.
The safety and tolerability of Coenzyme Q10 | 3 months
  Assess the safety and tolerability of Coenzyme Q10 supplementation in pediatric SLE patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The Pediatric Allergy, Immunology and Rheumatology Unit, Ain Shams University Hospitals., Cairo, Egypt